CLINICAL TRIAL: NCT01747109
Title: A Prospective, Multicenter, Randomized, Controlled, Parallel-group, Open Label Trial Evaluating Benefits of Nasal High Flow Therapy (HFT) in Preoxygenation Before Tracheal Intubation in Acute Hypoxemic Respiratory Failure
Brief Title: Benefits of Optiflow® Device for Preoxygenation Before Intubation in Acute Hypoxemic Respiratory Failure : The PREOXYFLOW Study
Acronym: PREOXYFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC12_0178
Record Dates: First submitted 2012-12-04; First posted 2012-12-11 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: Acute hypoxemic respiratory failure; Preoxygenation; Crash induction
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PREOXYFLOW (Experimental): Patients randomized in "PREOXYFLOW" group will received a four minutes preoxygenation period with Nasal High Flow Therapy (HFT) Optiflow ® (60 l/mn FIO2 = 1) before orotracheal intubation under laryngoscopy after crash induction
  Interventions: Device: PREOXYFLOW
- STANDARD FACE MASK (Active Comparator): Patients randomized in "STANDARD FACE MASK" group will received a four minutes preoxygenation period with a standard face mask (15 l/mn) before orotracheal intubation under laryngoscopy after crash induction. No specific trademark is requested by the protocol.
  Interventions: Procedure: STANDARD FACE MASK

INTERVENTIONS:
Device: PREOXYFLOW — Patients randomized in "PREOXYFLOW" group will received a four minutes preoxygenation period with Nasal High Flow Therapy (HFT) Optiflow ® (60 l/mn FIO2 = 1) before orotracheal intubation under laryngoscopy after crash induction
  Arms: PREOXYFLOW
Procedure: STANDARD FACE MASK — Patients randomized in "STANDARD FACE MASK" group will received a four minutes preoxygenation period with a standard face mask (15 l/mn) before orotracheal intubation under laryngoscopy after crash induction. Each hospital involved in this study will use the standard face mask as per its usual practice (no specific trademark requested by this protocol)
  Arms: STANDARD FACE MASK

SUMMARY:
Oro-tracheal intubation in intensive unit care(ICU) in acute hypoxemic respiratory failure after crash induction remains a critical event.

The aim of this study is to determine whether Nasal High Flow Therapy (HFT) Optiflow ® is more efficient than the face mask for preoxygenation before orotracheal intubation after crash induction in acute hypoxemic respiratory failure

DETAILED DESCRIPTION:
This study will be designed as followed : Patients will be randomized in 2 groups :"PREOXYFLOW" or "STANDARD FACE MASK".

Patients randomized in "PREOXYFLOW" group will received a four minutes preoxygenation period with Nasal High Flow Therapy (HFT) (60 l/mn FIO2 = 1) before orotracheal intubation under laryngoscopy after crash induction. Patients randomized in "STANDARD FACE MASK" group will received a four minutes preoxygenation period with standard face mask (15 l/mn) before orotracheal intubation under laryngoscopy after crash induction

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 years regardless of the gender
* Acute hypoxemic respiratory failure defined as :

Respiratory rate > 30/mn AND Hypoxemia with SpO2 <90% with oxygen supply > FiO2 0,5 AND PaO2/FiO2 <300 mmHg

Exclusion Criteria:

* Contraindication to oro-tracheal intubation
* Intubation without anesthetic delivery
* Intubation during cardiac arrest
* Asphyxia with immediate intubation needed
* Nasopharyngeal obstacle with contraindication to use Optiflow device
* Patients with a documented Cormack IV exposition before inclusion
* Protected adult
* Pregnancy
* Lack of consent
* Patient already enrolled in an other randomized study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
to determine whether Optiflow® used during the preoxygenation period before orotracheal intubation after crash induction is more efficient than standard face mask. | 4 minutes
  This outcome will be assessed from the beginning of the preoxygenation period to the end of orotracheal intubation by monitoring the pulse oxymetry

SECONDARY OUTCOMES:
Improvement of quality of preoxygenation | 4 minutes
Reduction in side effects incidence related to intubation | 1 hour
Reduction in Organ failure in the 5th day | at day 5
Reduction in morbi-mortality during the Intensive Care Unit stay. | until day 28 OR, if patient still in the intensive care unit (ICU) at Day 28, until discharge of ICU

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Nantes Universitary Hospital, medical intensive care unit, Nantes, Loire Atlantique
  - Angers Universitary Hospital, Angers
  - Brest Universitary Hospital, Brest
  - La Roche/Yon Hospital, La Roche/Yon
  - Montpellier University hospital, Montpellier
  - Nantes Universitary Hospital, surgical intensive care unit, Nantes

REFERENCES:
- [Derived] Vourc'h M, Asfar P, Volteau C, Bachoumas K, Clavieras N, Egreteau PY, Asehnoune K, Mercat A, Reignier J, Jaber S, Prat G, Roquilly A, Brule N, Villers D, Bretonniere C, Guitton C. High-flow nasal cannula oxygen during endotracheal intubation in hypoxemic patients: a randomized controlled clinical trial. Intensive Care Med. 2015 Sep;41(9):1538-48. doi: 10.1007/s00134-015-3796-z. Epub 2015 Apr 14. PMID 25869405